CLINICAL TRIAL: NCT07406646
Title: The Role of Monitoring of the Circulating and Urinary Exosomal miRNA for Prediction of Response to Treatment in Patients With Advanced Kidney Cancer
Brief Title: Circulating and Urinary Exosomal miRNA in Advanced Kidney Cancer (EXO-RENAL1)
Acronym: EXO-RENAL1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OI-EXO-RENAL1; ERID-KSOPKR-0083/2021 (Other: Clinical Research Unit, Institute of Oncology Ljubljana)
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Renal Cell Carcinoma; Advanced Kidney Cancer
Keywords: Exosomal miRNA; Circulating Biomarkers
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EXO-RENAL1 Cohort (Other): Patients with advanced renal cell carcinoma receiving standard-of-care systemic treatment (immune checkpoint inhibitors or targeted therapy) in the first-line or second-line setting. Circulating and urinary exosomal miRNA will be monitored during the first 16 weeks of treatment using blood and urine samples.
  Interventions: Other: Blood and Urine Sampling for Exosomal miRNA Analysis

INTERVENTIONS:
Other: Blood and Urine Sampling for Exosomal miRNA Analysis — Collection of peripheral blood and urine samples for analysis of circulating and urinary exosomal miRNA during the first 16 weeks of systemic treatment in patients with advanced renal cell carcinoma.

SUMMARY:
This prospective cohort study will investigate whether changes in circulating and urinary exosomal biomarkers (target exosomal miRNA) are associated with response to systemic treatment in patients with advanced renal cell carcinoma. Patients treated with immune checkpoint inhibitors or targeted therapies in the first-line or second-line setting will be included. Exosomal biomarker expression will be analyzed in blood and urine samples collected during the first 16 weeks of treatment. Treatment response will be assessed using standard radiological imaging. The study aims to determine whether changes in exosomal miRNA expression after treatment initiation can serve as predictive biomarkers of objective response in advanced kidney cancer.

DETAILED DESCRIPTION:
This is a prospective observational cohort study conducted at the Institute of Oncology Ljubljana. The study will evaluate the predictive value of circulating and urinary exosomal biomarkers (target exosomal miRNA) for response to systemic therapy in patients with advanced renal cell carcinoma.

Patients receiving immune checkpoint inhibitors or targeted therapy in the first-line or second-line treatment setting will be enrolled. The primary objective is to determine whether changes in the expression of selected exosomal miRNA in plasma after initiation of systemic treatment are associated with objective response to therapy. In addition, urinary exosomal miRNA will be evaluated as a potential predictive biomarker.

Blood and urine samples will be collected during the first 16 weeks of treatment. Each participant will provide four peripheral blood samples (10 mL each) and two urine samples (50 mL each). Radiological imaging will be performed as part of routine clinical follow-up to assess treatment response. The association between changes in exosomal miRNA expression and treatment outcomes will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (≥ 18 years).

Histologically confirmed advanced renal cell carcinoma.

Patients receiving systemic treatment with immune checkpoint inhibitors or targeted therapy in the first-line or second-line setting.

Ability to provide blood and urine samples according to the study protocol.

Signed informed consent.

Exclusion Criteria:

Patients unable to provide required biological samples.

Patients with missing clinical or imaging data required for treatment response assessment.

Any condition that, in the investigator's opinion, makes the patient unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Change in Plasma Exosomal miRNA Expression and Objective Response | During the first 16 weeks of treatment
  To determine whether changes in the expression of target plasma exosomal miRNA after initiation of systemic treatment are associated with objective response to treatment in patients with advanced renal cell carcinoma receiving immune checkpoint inhibitors or targeted therapy.

SECONDARY OUTCOMES:
Change in Urinary Exosomal miRNA Expression and Objective Response | During the first 16 weeks of treatment
  To determine whether changes in the expression of target urinary exosomal miRNA after initiation of systemic treatment are associated with objective response to treatment in patients with advanced renal cell carcinoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No